CLINICAL TRIAL: NCT05143944
Title: Audit of Management of First Stage of Labour in Assiut University Hospitals : a Quality Improvement Project
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Maksy, audit of management of first stage of labour in Assiut university hospitals : a quality improvement project, Assiut University
Other Study IDs: audit of first stage of labour
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nice clinical guidelines for intrapartum care for healthy women and babies: define gold standards in intrapartum care for healthy women and babies
- performance in the care provided to patients in periods of audit: measure performance in the care provided to the patients in the period of audit

SUMMARY:
auditing the current management of first stage of normal vaginal deliveries at Assiut university hospitals emergency obstetric care

DETAILED DESCRIPTION:
Clinical auditing is a quality improvement process that involves reviewing the delivery of healthcare to ensure the best practice is being carried out . it is agreed that caesarean section rates are above the nationally accepted in Egypt . This can be related to many factors and can be associated with risks to morbidities and mortalities

ELIGIBILITY:
Inclusion Criteria:

* term 37- 41 weeks primigravida single vertex presentation living fetus spontaneous onset no contraindications for vaginal delivary

Exclusion Criteria:

* women with associated co morbidities pre eclampsia and diabetes IUFD previous uterine scar intrauterine growth restriction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all women in reproductive age
Study Population: normal vaginal dellivary of primigravida
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
measure performance according to gold standers | BASELINE
  measure performance and adherence to gold standers during management of first stage of labour in assuit university hospitals

SECONDARY OUTCOMES:
introduction of NICE guidelines in practice | baseline
  introduction of NICE guidelines in management of first stage of labour in practice in assuit university hospitals